CLINICAL TRIAL: NCT00432055
Title: A Randomized Controlled Trial on Effects of Botulinum Toxin Type A in Adults With Cerebral Palsy
Brief Title: Effects of Botulinum Toxin Type A in Adults With Cerebral Palsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Johan K Stanghelle, Sunnaas Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20624503; EudraCTnumber: 2006-001427-19
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Cerebral Palsy
Keywords: Adult; Cerebral Palsy; Spastic contractures; Botulinum toxin type A
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Botox
  Interventions: Drug: Botulinum toxin type A (Botox)
- II (Placebo Comparator)
  Interventions: Drug: placebo (saline)

INTERVENTIONS:
Drug: Botulinum toxin type A (Botox)
  Arms: I
Drug: placebo (saline)
  Arms: II

SUMMARY:
The purpose of this project is to investigate if there is a significant difference in active joint range of motion, questionnaire on gait function and health related quality of life between patients randomized to treatment with Botulinum toxin type A and patients randomized to placebo treatment.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a constellation of symptoms and conditions defined as lifelong motor dysfunction resulting rom a non-progressive brain lesion occurring pre-, peri- or postnatal before the second year of life. CP consists of different aspect of motor disorder including spasticity, paresis, incoordination and dystonia

There is scarce knowledge about the association between spasticity, pain and physical function in the adult CP-population, and the systematic follow up of patients with CP typically ends at the age of eighteen. Frequently used intervention in spastic cerebral palsy for children with gait problems are injections with Botulinum toxin type A (Btx-A) in leg and thigh muscles, and three dimensional-gait analysis has become a standard procedure in treatment decision and evaluation.

Botulinum toxin A (Btx- A) is a highly effective treatment in the management of spasticity. The first reported success of use of Btx-A in children with cerebral palsy was made in 1993 by Koman et al. Subsequently, randomized controlled studies on children with spastic type of cerebral palsy has documented that Btx-A is effective and safe in the management of muscle spasticity in children with CP. There is an implicit, and as of yet, unproven assumption that there is no indication for this treatment in the adult CP-population.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral spastic CP
* Modified Ashworth Scale (MAS) ≥ 2 in ankle- or knee joint muscles.
* ≥ 18 year of age, ≤ 65 year of age
* Ambulant without walking aids minimum 10 metres in functional equines and/or with pathological knee extension or flexion pattern.

Exclusion Criteria:

* Cognitive impairment.
* No spasticity (MAS < 2 )
* < 18 year of age
* Not ambulant without walking aids
* Pregnant or planning pregnancy
* Btx-A treatment last 6 months
* Orthopedic surgery lower extremity last 18 months
* Obvious skeletal/joint deformity where orthopedic surgery is indicated
* Other diseases which can affect level of function (rheumatoid or neurological )
* New treatment the past four weeks which affect the musculoskeletal system (pain killers, physical therapy, acupuncture)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Ankle sagittal kinematic with corresponding knee and hip data (3D-gait analysis) | 8 week
Summary measure of health related quality of life (SF-36) | 8 week , 16 week

SECONDARY OUTCOMES:
Stiffness/spasticity according to VAS | 8 week, 16 week
Questionnaire gait function | 8 week, 16 week
Spasticity in ankle, knee and hip according to Modified Ashworth Scale | 8 week,
3D-gait data (Kinetics,Temporospatial (stride length, velocity) | 8 week
Global Scale | 8 week, 16 week
Timed Up and Go | 8 week
6 minutes walking test | 8 week
Registrations of sample characteristics | 0 week
Registration of adverse reactions | 8 week, 16 week
Pain according to VAS | 8 week, 16 week

CONTACTS AND LOCATIONS:
Overall Officials: Johan K Stanghelle, Professor MD, Study Chair — Research Departement, Sunnaas Rehabilitation Hospital
Locations (1):
- Sunnaas Rehabilitation Hospital, Bjoernemyr, Nesoddtangen, Norway